CLINICAL TRIAL: NCT06533943
Title: Engaging in Physical Activity Carried Out in a Blue-green Space to Improve Health, Quality of Life and Physical Performance Among the Population: the "Parco Del Mare" Study Protocol
Brief Title: Blue-green Space Physical Activity: the "Parco Del Mare" Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Sofia Marini, Researcher, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0121439
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy Adults; Natural Outdoor Environment; Health Promotion
Keywords: blue-green space setting; physical activity intervention; outdoor exercise; public health
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group (EG) undergo the exercise program designed for the purpose of the study. The outdoor sessions will be carried out in groups (2 sessions per week, lasting 1 hour each one) and administered by trainers with a master's degree in Science and Technique of Preventive and Adapted Physical Activity (kinesiologists).
  Interventions: Other: Exercise program
- Control Group (No Intervention): The control group (CG) will be asked to abstain from structured exercise or training, limiting their physical effort to activities needed for daily life.

INTERVENTIONS:
Other: Exercise program — Each intervention session is divided into three different parts according to the specific aim such as warm-up (about 15 minutes) at the beginning, main exercises (about 30 minutes), and stretching and relaxation (about 15 minutes) at the end.
  Arms: Experimental group

SUMMARY:
This study protocol, describe the innovative study intervention which will be performed in a green-blue space in Italy in order to investigate on the improvements in wellbeing following participation in the study. This will be significant because it will provide evidence on the effectiveness of the supervised physical activities carried out in green-blue space in improving health, quality of life, physical performance, anthropometric outcomes and physiological parameters in adults, indicating the reasonableness for public health authorities to developing such activities.

DETAILED DESCRIPTION:
The aim of the "Parco del Mare" pilot study is to evaluate the feasibility and the effects of a moderate-intensity exercise program carried out in a green-blue space, on health outcomes such as quality of life and physical performance. Healthy adults with no contraindication to practice physical activity will be recruited and divided into two groups: the experimental group involved in the exercise sessions performed twice a week for 6-months, while the control group received no intervention. Validated tests and questionnaires will be used to detect health parameters at baseline (T0) and follow-up (T1). The investigators expected the intervention carried out in the Parco del Mare setting to be feasible and effective in improving health parameters, quality of life and physical performance in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult population aged >18 years old
* Resident in Rimini

Exclusion Criteria:

* Any alterations in communication skills and/or sensory functions so severe as to make it impossible to understand and/or execute the instructions given by the trainer (dementia, aphasia, blindness, deafness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
12-Item Short Form Survey (SF-12) | through study completion, an average of 1 year
  Quality of Life measurement (higher scores indicate better physical and mental components)

CONTACTS AND LOCATIONS:
Locations (1):
- Parco del Mare, Rimini, Rimini, Italy